CLINICAL TRIAL: NCT03566836
Title: Atrial Fibrillation Detection Using Garmin Wearable Technology
Acronym: GARMIN AF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Garmin International (Industry)
Responsible Party: Sponsor
Other Study IDs: STUDY00142473
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Atrial Fibrillation
Keywords: Smart Watch; Garmin; Wearable; Cardioversion
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- AF Detection: Participants will be asked to wear the Garmin smart watch and Garmin chest band. Both are commercially available. The devices will collect information about heart rates before and after a cardioversion procedure.
  Interventions: Device: Garmin Smart Watch; Device: Garmin Chest Band

INTERVENTIONS:
Device: Garmin Smart Watch — Garmin Smart Watch
Device: Garmin Chest Band — Garmin Chest Band

SUMMARY:
The purpose of this study is to evaluate the feasibility of detecting atrial fibrillation (AF) in patients with AF using a wearable wrist device/smart watch.

DETAILED DESCRIPTION:
Even though AF is common and associated with increased risk of stroke, quite often it goes undetected until late in the course of the condition. If AF can be detected with simpler tools like a smart watch, it would enable providers to identify patients with AF much earlier in the course of the condition (even before being seen by a physician) and hopefully be able to prevent stroke. This study is being done to identify a technology that can likely identify AF using a smart watch.

ELIGIBILITY:
Inclusion Criteria:

* All patients with AF scheduled to undergo electrical cardioversion at the University of Kansas Health System

Exclusion Criteria:

* Patients with no detectable PPG
* Hemodynamically unstable patients
* Patients who cannot give informed consent
* Patients with tattoos on the wrists

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are receiving care from the University of Kansas Health System.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-06-19 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of Garmin wearable device in detecting AF | Visit 1
  PPG samples collected from Garmin wearable will be evaluated and calculated by Garmin custom

CONTACTS AND LOCATIONS:
Overall Officials: Yeruva Madhu Reddy, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided